CLINICAL TRIAL: NCT05843006
Title: SWEAT Analysis for Predicting Patient Outcome After HEART Attack
Brief Title: Sweat Analysis as Prognosticator After Heart Attack
Acronym: SWEATHEART
Status: Completed | Type: Observational
Sponsor: Region Örebro County (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 274564
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2022-03

CONDITIONS: Acute Myocardial Infarction
Keywords: Sweat analysis; Myocardial reperfusion injury; Personalized patient monitoring; Acute myocardial infarction; Upregulated sympathetic nervous system; Inflammation
MeSH Terms: conditions — Myocardial Reperfusion Injury; Inflammation | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples With DNA — Sweat and venous blood samples for analysis and storage in a biobank in Örebro for potential future analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STEMI + PCI: 18 subjects referred for coronary angiography/PCI due to ST-segment elevation myocardial infarction (STEMI)
  Interventions: Diagnostic Test: Examination and analysis of sweat and blood samples at baseline and at follow up
- Diagnostic coronary angiography without a resulting intervention (PCI): 6 subjects undergoing a diagnostic coronary angiography without a resulting intervention (PCI)
  Interventions: Diagnostic Test: Examination and analysis of sweat and blood samples at baseline

INTERVENTIONS:
Diagnostic Test: Examination and analysis of sweat and blood samples at baseline and at follow up — Subjects will be assessed at baseline (as inpatients) and at 4-6 weeks at follow-up as outpatients according to standard operating procedures. Sweat samples will be collected using the CE certified Macroduct Sweat Collector and inflammatory parameters measured. Venous blood will be drawn and inflammatory parameters, Troponin-I and nt-proBNP measured. Further examinations include measurement of left ventricular ejection fraction by echocardiography at baseline and blood pressure, heart rate, risk scores and health information will be collected at baseline and follow up.
  Groups: STEMI + PCI
Diagnostic Test: Examination and analysis of sweat and blood samples at baseline — Sweat samples will be collected using the CE certified Macroduct Sweat Collector and inflammatory parameters measured. Venous blood will be drawn and inflammatory parameters, Troponin-I and nt-proBNP measured. Blood pressure, heart rate, risk scores and health information will collected.
  Groups: Diagnostic coronary angiography without a resulting intervention (PCI)

SUMMARY:
This study characterizes non-invasive body inflammation response in sweat and blood of patients suffering from acute myocardial infarction and explores the potential of non-invasive sweat analysis a an innovative approach for predicting patient outcome.

DETAILED DESCRIPTION:
Background:

Different risk scores exist for predicting patient outcome after acute coronary syndrome and percutaneous coronary intervention (PCI). This is of importance to optimize post interventional patient management as well as treatment and to reduce the risks of re-hospitalization and mortality. ST-elevation myocardial infarction (STEMI) has been associated with an instant upregulation of the sympathetic nervous system leading to adrenergic stimulation and immune system activation in different organs such as the heart and skin. In skin, sympathetic fibers travel together, appear as single nerve fibers in the dermis as well as in the epidermis, and activate inflammation by norepinephrine secretion. Further, STEMI has been associated with increased sweating during the acute phase. In an unpublished pilot trial, we detected a broad panel of inflammation markers in sweat (such as MCP-1, TGFβ, uPa, TRAIL) of healthy volunteers. Sweat immunologic marker analysis is an interesting and novel approach for assessment of sympathetic activation and inflammation.

Objective and methods:

Our primary objective is to assess a non-invasive body inflammation response in sweat and blood of patients suffering from STEMI after PCI (+4h) and at outpatient follow up (±4-6 weeks). Body inflammation marker concentrations in sweat and blood will be set into context to cardiovascular risk factors, GRACE and TIMI STEMI scores, door-to-balloon time, length of hospital stay , left ventricular ejection fraction, peak troponin-I, and NT-proBNP concentrations to investigate the STEMI/PCI - sympathetic nervous system - inflammation axis. A total of 18 subjects with STEMI and 6 patients undergoing diagnostic coronary angiography without PCI will be recruited in a clinical, single-center pilot study at Örebro University Hospital. Sweat will be collected using the CE certified Macroduct Collecting System and blood samples will be taken. Analysis will be performed with Olink proteomic analysis.

Clinical relevance:

STEMI and subsequent reperfusion are associated with an increase in inflammatory response. Myocardial reperfusion injury contributes significant to myocardial injury after STEMI. Adequate patient monitoring and therapy after PCI is essential to preserve cardiac function, prevent re-hospitalization, heart failure and death.

Prospects:

Biomarkers can be collected by smart biosensors and may provide novel longitudinal insights into health and disease. On-skin sweat analysis using wearable devices are increasingly available and will allow collection of non-invasive and patient-centered molecular health information in the future. This may help to investigate a better understanding of sympathetic nervous system upregulation after STEMI/PCI.

ELIGIBILITY:
Inclusion Criteria:

Study participants will be recruited among subjects referred to Hospital for coronary angiography/PCI due to ST-segment elevation myocardial infarction (STEMI) or diagnostic coronary angiography.

Subjects with a diagnosis of STEMI as defined by chest pain suggestive for myocardial ischemia for at least 30 minutes before hospital admission, time from onset of symptoms of less than 24 hours, and an ECG with new ST-segment elevation in two or more contiguous leads of ≥0.2 mV in leads V2-V3 and/or ≥0.1 mV in other leads or a probable new-onset left bundle branch block

Or:

Subjects undergoing a diagnostic coronary angiography without a resulting intervention (PCI)

and:

Written informed consent

Exclusion Criteria:

* Emergency coronary artery bypass grafting
* On immunosuppression pharmacotherapy
* Pacemaker patients

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited among patients referred to Örebro University Hospital a tertiary teaching hospital and regional acute care hospital.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Inflammation panels in sweat and blood correlated to clinical outcome | 6 weeks
  The primary result is detection of inflammation markers in sweat and blood samples in patients with STEMI and PCI. Inflammation markers will be correlated to clinical outcome. Clinical endpoints will be assessed in all patients included in the study using data from the Swedish Web System for Enhancement and Development of Evidence-based Care in Heart Disease Evaluated According to Recommended Therapies (SWEDEHEART) registry - death, new AMI and new, unplanned revascularization. Assessment is exploratory only.

SECONDARY OUTCOMES:
Comparing inflammation panels of patients with coronary angiography without any need for an intervention | 6 weeks
  Secondary results are detection of inflammation markers in sweat and blood of patients with coronary angiography but no need for intervention and compared to patients with STEMI and PCI. Clinical endpoints will be assessed as described for the primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Ole Fröbert, MD, PhD, Study Chair — Department of Cardiology, Örebro University Hospital and Örebro University
Locations (1):
- Department of cardiology, Örebro, Sweden

REFERENCES:
- [Derived] Bjorkenheim A, Sunnefeldt E, Finke K, Smith DR, Frobert O, Brasier N. Biomarkers of inflammation in sweat after myocardial infarction. Sci Rep. 2025 Feb 15;15(1):5564. doi: 10.1038/s41598-025-90240-8. PMID 39955425